CLINICAL TRIAL: NCT00365521
Title: Prophylactic Photodynamic Therapy to Organ Transplant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: KF-01-314759
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Organ Transplants
Keywords: Organ transplant patients receiving immunosuppressive therapy
MeSH Terms: interventions — Photochemotherapy

INTERVENTIONS:
Procedure: Photodynamic Therapy

SUMMARY:
To evaluate a possible prophylactic efficacy of photodynamic therapy on the incidence of non-melanoma skin cancer, actinic keratoses, warts and keratoses in recently organ transplanted recipients.

ELIGIBILITY:
Inclusion Criteria:

* Organ transplant recipients.
* Age 40 years or older.

Exclusion Criteria:

* Patients younger than 40 years and older than 70 years.
* Clinical signs of skin cancer, actinic keratoses or warts at the time of inclusion.
* Previous photodynamic therapy to the skin areas investigated.
* Pregnancy or breast feeding patients.
* Patients with porphyria.
* Patients with a tendency to produce hypertrophic scars or keloids.
* Patients with known allergy to Metvix.
* Patients who are not considered able to follow the treatment protocol (e.g. severely alcoholic patients, dementia patients, mentally ill patients etc.).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-04

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, MD, PhD, DrMedSci, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark